CLINICAL TRIAL: NCT07089823
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of YP05002 in Healthy Participants
Brief Title: A Study of YP05002 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yaopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YP05002-001
Record Dates: First submitted 2025-07-25; First posted 2025-07-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental): SAD dose 1
  Interventions: Drug: YP05002; Other: Placebo
- SAD Cohort 2 (Experimental): SAD dose 2
  Interventions: Drug: YP05002; Other: Placebo
- SAD Cohort 3 (Experimental): SAD dose 3
  Interventions: Drug: YP05002; Other: Placebo
- SAD Cohort 4 (Experimental): SAD dose 4
  Interventions: Drug: YP05002; Other: Placebo
- SAD Cohort 5 (Experimental): SAD dose 5
  Interventions: Drug: YP05002; Other: Placebo
- MAD Cohort 1 (Experimental): MAD dose 1
  Interventions: Drug: YP05002; Other: Placebo
- MAD Cohort 2 (Experimental): MAD dose 2
  Interventions: Drug: YP05002; Other: Placebo
- MAD Cohort 3 (Experimental): MAD dose 3
  Interventions: Drug: YP05002; Other: Placebo

INTERVENTIONS:
Drug: YP05002 — Tablet, QD
Other: Placebo — Tablet, QD

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled, single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, efficacy, food effect of YP05002 Tablets in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
2. Healthy male and female participants aged 18-65 years (both inclusive).No restrictions on race.
3. In good health as determined by the Investigator, with no clinically significant findings from medical/psychiatric history, physical examination, 12-lead ECG, vital signs measurements, clinical laboratory evaluations.

Exclusion Criteria:

1. Have evidence of any clinically significant active or chronic disease.
2. Histories of using drug that affect drug absorption, distribution, metabolism, or excretion within 14 days or within 5-half-life prior to the first dose (whichever is longer); gastrointestinal disorders with impaired gastric emptying; or prolonged use of medications that directly modulate gastrointestinal motility.
3. Had clinically relevant acute or chronic medical conditions or diseases that would pose a risk to participant's safety or interfere with the study assessments, as determined by the Investigator.
4. Any malignancy (except basal cell carcinoma and squamous cell carcinoma of the skin) in the previous 5 years.
5. Diagnosis of any type of pancreatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of adverse events (AEs), serious adverse events (SAEs) in each dose group during the safety observation period (SAD) | Up to Day 14
Number and percentage of adverse events (AEs), serious adverse events (SAEs) in each dose group during the safety observation period (MAD) | Up to Day 41

SECONDARY OUTCOMES:
Cmax of YP05002 (SAD) | Up to Day 14
  PK parameters of YP05002
Cmax of YP05002 (MAD) | Up to Day 41
  PK parameters of YP05002

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne Clinic, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No